CLINICAL TRIAL: NCT02031549
Title: Prospective Observational Correlation of Sperm Assay Results With Blastocyst Formation
Status: Completed | Type: Observational
Sponsor: Bruce Shapiro M.D. (Industry)
Responsible Party: Sponsor-Investigator, Bruce Shapiro M.D., Medical Director, Fertility Center of Las Vegas
Organization: Fertility Center of Las Vegas (Industry)
Other Study IDs: SAIRB-13-0038
Record Dates: First submitted 2014-01-07; First posted 2014-01-09 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-03

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- SpermComet Assay: All study subjects will have their surplus sperm analyzed for DNA fragmentation with the SpermComet assay.
  Interventions: Other: SpermComet assay

INTERVENTIONS:
Other: SpermComet assay — Measurement of DNA fragmentation in samples of surplus sperm (diagnostic, not an intervention).

SUMMARY:
We will investigate potential correlation between SpermComet DNA fragmentation assay results and IVF cycle outcome.

DETAILED DESCRIPTION:
A "SpermComet" assay will be used to characterize DNA fragmentation of surplus sperm samples remaining after in vitro fertilization (IVF) cycles. We will investigate potential correlation between these assay results and the outcomes of IVF cycles that used those sperm samples.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing IVF
* Surplus sperm available after oocyte insemination
* Consented

Exclusion Criteria:

* Surgical sperm extraction
* Use of donated sperm or oocytes
* No minors may participate

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Couples who undergoing IVF treatment who have surplus sperm available after oocyte insemination.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2014-01; Primary Completion 2014-02 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Blastulation rate | 6 days
  The proportion of oocytes and of fertilized oocytes that form blastocysts.

SECONDARY OUTCOMES:
Fertilization rate | 1 day
  Proportion of inseminated oocytes that form exactly two pronuclei.
Embryo grade | 6 days
  Grade and measurements of blastocysts that form.

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Shapiro, MD, PhD, Principal Investigator — Fertility Center of Las Vegas
Locations (1):
- Fertility Center of Las Vegas, Las Vegas, Nevada, United States